CLINICAL TRIAL: NCT01107730
Title: Randomized Double Blind Study of Administration of Vitamin C for Prophylaxis of Post-operative Atrial Fibrillation in On-pump Cardiac Surgery Procedures
Brief Title: Vitamin C for Prophylaxis of Post-operative Atrial Fibrillation in On-pump Cardiac Surgery Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Polymeropoulos Evangelos, Dr, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 268/27-07-09
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Cardiac valve repair; Aneurysm repair; CABG; On-pump; Cardiac surgery; Vitamin C
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ascorbic Acid; Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- L-Carnitine (Active Comparator): L-Carnitine intravenously (2 gr/day [1grX2] for 2 days prior to surgery, and postoperatively for 4 days
  Interventions: Drug: L-Carnitine
- Vitamin C (Active Comparator): VitC intravenously (2g/day [500mgX4] for 2 days prior to surgery, and postoperatively for 4 days
  Interventions: Drug: Vitamin C
- Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C — VitC intravenously (2g/day [500mgX4] for 2 days prior to surgery, and postoperatively for 4 days
  Arms: Vitamin C
Drug: L-Carnitine — L-Carnitine intravenously (2 gr/day [1grX2] for 2 days prior to surgery, and postoperatively for 4 days
  Arms: L-Carnitine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether vitamin C is effective in the prophylaxis of post-operative atrial fibrillation in on-pump cardiac surgery

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the single most common post-operative complication after on-pump cardiac surgery, ranging from roughly 25% in CABG procedures, up to 65% in valve replacement procedures. The presence of AF in cardiac surgery patients doubles the morbidity amongst these patients, as well as raising the mortality rates. VitC is an electron donor for a number of enzymatic systems, reducing potentially harmful free radicals. In post-procedural AF, there is increased peroxynitrite concentration, which is a target for vitamin C. A randomized, double blind study will be conducted in order to establish the efficiency of vitamin C as prophylaxis for postoperative AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing on-pump cardiac surgery

Exclusion Criteria:

* Off-pump cardiac surgery procedure
* AF before the procedure
* Recent infection and/or infectious endocarditis
* Presence of neoplasia
* Chronic renal failure with creatinine>2.3 mg/dl
* Hepatic failure
* Autoimmune disease and/or disease that brings about a systematic inflammatory response
* Thyroid disease
* Systematic use of supplements that contain vitC or carnitine
* The use of NSAIDs other than aspirin for a time period up to one month before the procedure

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Toumpoulis, MD, Study Chair — University of Athens Medical School, Attikon Hospital, Cardiology Department
Locations (1):
- University General Hospital Attikon, Athens, Greece

REFERENCES:
- [Result] Rodrigo R, Vinay J, Castillo R, Cereceda M, Asenjo R, Zamorano J, Araya J, Castillo-Koch R, Espinoza J, Larrain E. Use of vitamins C and E as a prophylactic therapy to prevent postoperative atrial fibrillation. Int J Cardiol. 2010 Feb 4;138(3):221-8. doi: 10.1016/j.ijcard.2009.04.043. Epub 2009 May 15. PMID 19446899

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | L-Carnitine | Vitamin C | Placebo
Started | 11 | 11 | 11
Completed | 11 | 11 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- L-Carnitine: Carnitine 2 days preoperatively and 4 days postoperatively
- Vitamin C: Vitamin C 2 days preoperatively and 4 days postoperatively
- Total: Total of all reporting groups
Arm/Group | L-Carnitine | Vitamin C | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 11 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 5 | 14
  >=65 years | 8 | 5 | 6 | 19
Age, Continuous [Median (Full Range); unit: years] | 75 [42 to 85] | 64 [41 to 79] | 65 [44 to 87] | 66 [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 7 | 7 | 6 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 11 | 11 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 11 | 11 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Atrial Fibrillation
Description: The incidence of postoperative atrial fibrillation in cardiac surgery patients, using 2 different prophylaxis regimens with vitamin C, as compared to placebo.
Time Frame: Within the first 30 days (plus or minus 3 days)
Measure: Number; unit: participants
Arm/Group | L-Carnitine | Vitamin C | Placebo
Number analyzed (Participants) | 11 | 11 | 11
participants | 5 | 4 | 5

ADVERSE EVENTS:
Groups:
- L-Carnitine: Carnitine 2 days preoperatively and 4 days postoperatively
  Carnitine: Carnitine 2 days preoperatively and 4 days postoperatively
- Vitamin C: Vitamin C 2 days preoperatively and 4 days postoperatively
  Vitamin C: Vitamin C 2 days preoperatively and 4 days postoperatively
Arm/Group | L-Carnitine | Vitamin C | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No